CLINICAL TRIAL: NCT00662948
Title: Open Study in Phase II to Evaluate Efficacy of Initial R-CHOP Combination in Folicular Lymphoma no Treated Previously. Consolidation w Ith One Dose of 90Y Ibritumomab Tiuxetan (Zevalin®) Versus Maintenance Treatment With Rituximab (MabThera®)
Brief Title: ZAR2007: R-CHOP in Folicular Lymphoma Patients no Treated Previously. Consolidation With 90Y Ibritumomab Tiuxetan (Zevalin®) Versus Maintenance Treatment With Rituximab (MabThera®)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Collaborators: GELCAB (Other); Grupo Español de Linfomas y Transplante Autólogo de Médula Ósea (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZAR2007
Record Dates: First submitted 2008-04-08; First posted 2008-04-21 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Lymphoma
Keywords: Folicular Lymphoma; Consolidation; Maintenance
MeSH Terms: conditions — Lymphoma | interventions — Rituximab; ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Consolidation with one dose of 90Y Ibritumomab tiuxetan (Zevalin®) 0,4 mCi/Kg
  Interventions: Drug: Ibritumomab tiuxetan
- B (Active Comparator): Maintenance with 375 mg/m2 of Rituximab every 8 weeks during 24 months
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — 375 mg/m2 every 8 weeks during 24 months
  Arms: B
Drug: Ibritumomab tiuxetan — One dose of 90Y Ibritumomab tiuxetan, 0,4 mCi/Kg
  Arms: A

SUMMARY:
After conventional induction treatment with R-CHOP (Rituximab, cyclophosphamide, adriamycin, vincristine and prednisone) the patients are randomized to:

A: Consolidation with one dose of 90Y Ibritumomab tiuxetan (Zevalin®) 0,4 mCi/Kg

B: Maintenance with 375 mg/m2 of Rituximab every 8 weeks during 24 months

DETAILED DESCRIPTION:
The study will evaluate the benefit of consolidation treatment with 90Y Ibritumomab tiuxetan (Zevalin®) or maintenance with rituximab (MabThera®) in terms of progression free survival, after induction with chemotherapy and rituximab in folicular lymphoma patients no treated previously.

The other aims are, evaluate the global survival, event free survival, time until next treatment, response rate after consolidation or maintenance treatment, quality of life, security of two branches and relation cost-efectivity

ELIGIBILITY:
Inclusion Criteria:

* Folicular Lymphoma CD20-positive, grade 1, 2 or 3a, confirmed in previous 4 months.
* Patients no treated previously.
* Ann Arbor Stage II, III o IV.
* Symptoms or signes wich indicate necesary treatment (GELF criteria):

  * Ganglionar or extraganglionar mass
  * B Symptoms
  * LDH or B2-microglobuline increased
  * 3 ganglionar territory afected (> 3 cm)
  * Esplenomegalia
  * Compresive syndrome
  * Pleural/peritoneal effusion
  * Secondary medular insufiency due to infiltration
* Age> 18 years and <75 years.
* ECOG < 2
* Adecuate hematological function: Hemoglobin > 8,0 g/dl (5,0 mmol/L); RAN >1,5 x 109/L; platelets > 100 x 109/L
* No pregnant women. Women and man should use an appropiate anticonceptive method during the study and one year after
* Informed consent

Exclusion Criteria:

* Transformation in high grade lymphoma
* FL grade 3b.
* Skin or gastro-intestinal primary lymphoma
* History of CNS diseases ( or CNS lymphoma)
* Previous treatment
* Regulary treatment with corticosteroids (permited < 20 mg/day prednisone or equivalent).
* Previous cancer diseases
* Major surgery in 28 days before inclusion in study.
* Creatinine > 2,0 mg/dl (197 mmol/L)
* Bilirubin > 2,0 mg/dl (34 mmol/L), AST (SGOT) > 3 x upper normal limit.
* HIV infection or active infection VHB o VHC < 4 weeks before inclusion.
* Other complicated diseases

Criteria investigador:

* Life expectancy < 6 months.
* Hipersensibility to Ibritumomab tiuxetan, rituximab, other murines proteins or any excipients.
* Treatment in other experimental study in previous 30 days
* Any medical o psicologycal condition that can modify the capacity to give the consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2008-12 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 2 years

SECONDARY OUTCOMES:
Saffetty of two arms | 2 years
Quality of life | 7 years
Global survival | 7 years
Event free survival | 7 years
Response rate in two arms | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Canales Miguel, Dr, Study Chair — Hospital La Paz; Lopez-Guillermo Armando, Dr, Study Chair — Hospital Clinic of Barcelona; Tomas Jose Francisco, Dr, Study Chair — MD Anderson- Madrid
Locations (21):
- Spain (21):
  - Hospital Juan Canalejo, A Coruña
  - Hospital de Alcorcón, Alcorcón
  - Hospital germans Trias i Pujol, Badalona
  - Hospital Clínic, Barcelona
  - Hospital de la santa Creu i Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Doce de Octubre, Madrid
  - Hospital La Paz, Madrid
  - Hospital Ramón y Cajal, Madrid
  - MD Anderson, Madrid
  - Hospital Virgen de la Arrixaca, Murcia
  - Hospital son Dureta, Palma de Mallorca
  - Hospital Clínico, Salamanca
  - Hospital de Donostia, San Sebastián
  - Hoaspital Marqués de Valdecilla, Santander
  - Hospital Clínico Universitario, Santiago de Compostela
  - Hospital Clínico, Valencia
  - Hospital Dr Pesset, Valencia
  - Hospital General, Valencia
  - Hospital La Fe, Valencia

REFERENCES:
- [Derived] Lopez-Guillermo A, Canales MA, Dlouhy I, Mercadal S, Briones J, Martin Garcia-Sancho A, Sancho JM, Moraleda JM, Terol MJ, Salar A, Palomera L, Gardella S, Jarque I, Ferrer S, Bargay J, Lopez A, Panizo C, Muntanola A, Montalban C, Conde E, Hernandez MT, Soler A, Garcia Marco JA, Deben G, Marin J, Tomas JF; PETHEMA/GELTAMO/GELCAB Spanish Intergroup. A randomized phase II study comparing consolidation with a single dose of 90Y ibritumomab tiuxetan vs. maintenance with rituximab for two years in patients with newly diagnosed follicular lymphoma responding to R-CHOP. Long-term follow-up results. Leuk Lymphoma. 2022 Jan;63(1):93-100. doi: 10.1080/10428194.2021.1971216. Epub 2021 Aug 30. PMID 34459702
- See also: spanish hematology association — http://aehh.org